CLINICAL TRIAL: NCT02029534
Title: Intensive Statin Therapy Effect on Incidence of Post-Operative Atrial Fibrillation
Brief Title: Intensive Statin Therapy Effect on Post-Operative Atrial Fibrillation (POAF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-16729
Record Dates: First submitted 2013-08-16; First posted 2014-01-08 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Cardiothoracic Surgery; Post-operative Atrial Fibrillation
Keywords: post-operative atrial fibrillation; POAF; A-Fib
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin 20 mg (Active Comparator): atorvastatin 20 mg daily 2 to 7 days prior to surgery and up to 7 post surgery
  Interventions: Drug: Atorvastatin 20 mg
- Atorvastatin 80 mg (Experimental): atorvastatin 80 mg daily 2 to 7 days prior to surgery and up to7 days post surgery
  Interventions: Drug: Atorvastatin 80 mg

INTERVENTIONS:
Drug: Atorvastatin 20 mg
  Other Names: Lipitor
  Arms: Atorvastatin 20 mg
Drug: Atorvastatin 80 mg
  Other Names: Lipitor
  Arms: Atorvastatin 80 mg

SUMMARY:
This study will compare the effects of 20 mg of atorvastatin to 80 mg of atorvastatin for the prevention of atrial fibrillation after cardiothoracic surgery. The study hypothesis is that 80 mg of atorvastatin will be more effective at preventing atrial fibrillation compared to 20 mg.

DETAILED DESCRIPTION:
This is a randomized, double-blind comparison of two doses of atorvastatin for prevention of post-operative atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or older
* Undergoing elective cardiothoracic surgery

Exclusion Criteria:

* Emergency cardiothoracic surgery
* History of permanent atrial fibrillation
* Acute coronary syndrome within 7 days
* Antiarrhythmic drug use in the past 3 months
* Receiving maximal tolerated dose of statin therapy
* Receiving fibrate therapy
* History of statin intolerance
* Significant liver impairment (aspartate aminotransferase/alanine aminotransferase(AST/ALT)>2x ULN)
* Serum Creatinine > 3 mg/dl
* Pregnancy or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of atrial fibrillation by hospital discharge | Hospital discharge, an expected 5-7 days
  Occurrence of atrial fibrillation, defined as a new diagnosis of atrial fibrillation that lasts at least 5 minutes based on telemetry or 12 lead ECG readings.

SECONDARY OUTCOMES:
Length of hospital stay | Hospital discharge, an expected 5-7 days
Incidence of major adverse cardiac and cardiovascular events (MACCE) at 30 days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Smer, MBBCh, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States